CLINICAL TRIAL: NCT04060849
Title: Prevention of Respiratory Viruses Using Nozin in Stem Cell Transplant Recipients (PREV-NOSE Study)
Brief Title: Nozin in Preventing Respiratory Viral Infections in Patients Undergoing Stem Cell Transplant, PREV-NOSE STUDY
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was closed to accrual according to the Fred Hutch/University of Washington/Seattle Children's Consortium low accrual institutional policy.
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: Global Life Technologies Corp. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RG1004525; NCI-2019-05159 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10087 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2019-08-14; First posted 2019-08-19 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Hematopoietic and Lymphoid Cell Neoplasm; Malignant Solid Neoplasm; Solid Neoplasm
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Practice Guidelines as Topic; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (Nozin) (Experimental): Beginning 7 days prior to transplant, patients receive Nozin via nasal single-use popswabs or single-use cotton tipped applicators and swab the inside of their nose BID up to 100 days after transplant.
  Interventions: Drug: Nozin
- Arm II (standard of care) (Active Comparator): Patients receive standard of care.
  Interventions: Other: Best Practice

INTERVENTIONS:
Drug: Nozin — Given via nasal single-use popswabs or single-use cotton tipped applicators
  Other Names: Ethanol-based Intranasal Solution; Ethanol-based Nasal Sanitizer; Ethanol-containing Nasal Solution
  Arms: Arm I (Nozin)
Other: Best Practice — Receive standard of care
  Other Names: standard of care; standard therapy
  Arms: Arm II (standard of care)

SUMMARY:
This phase I trial studies the side effects of Nozin in preventing respiratory viral infections in patients undergoing stem cell transplant. Nozin is a non-antibiotic, alcohol-based nasal sanitizer used in hospitals to prevent spread of bacterial infections and may also prevent community acquired respiratory virus infection in stem cell transplant recipients.

DETAILED DESCRIPTION:
OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Beginning 7 days prior to transplant, patients receive Nozin via nasal single-use popswabs or single-use cotton tipped applicators and swab the inside of their nose two times daily (BID) up to 100 days after transplant.

ARM II: Patients receive standard of care.

After completion of study, patients are followed up every week for 6 weeks and then every alternate week until day 100.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing allogeneic hematopoietic transplant for malignant or non-malignant disease
* English speaking
* Capable of providing informed consent
* Planned to receive follow-up at the transplant site for the first 100 days post transplantation
* Subjects who the investigator believes can and will comply with the study protocol

Exclusion Criteria:

* Documented respiratory viral infection in the two weeks prior to enrollment
* Current or planned use of any prophylactic antiviral therapy, antibody treatments, or other agents targeting the prevention of respiratory viruses (i.e. oseltamivir, ribavirin, amantadine)
* Known allergy to study drug components (jojoba, orange oil, coconut oil, lauric acid, benzalkonium chloride, vitamin E)
* Receiving oxygen supplementation at time of enrollment
* Active mucositis at time of enrollment
* Ongoing irritation or active infection of the squamous epithelial cell skin involving the nose or nasal vestibule
* Daily use of nasal decontamination products or other nasal medications (e.g. nasal steroids)
* Unable to complete study procedures (e.g. nasal swab self-testing)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-09-03 (Actual); Primary Completion 2020-04-12 (Actual); Study Completion 2020-04-12 (Actual)

PRIMARY OUTCOMES:
Tolerability of Nozin | Up to 100 days post-transplant
  Will measure and describe reasons for dropout, defined as failure to complete the study to day 100 for any reason. Among participants in the study product arm, reasons for dropout will be classified as either directly related to the product or due to other reasons. Will estimate the proportion of participants who exit the study for reasons directly related to the study product with a precision of +/- 20% (95% confidence interval) to inform tolerability of study product for future studies. Will compare dropout for any reason between treatment arms using Fisher's exact test.
Incidence of adverse events (AEs) | Up to 100 days post-transplant
  AEs will be graded in severity according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0. All adverse events will be continually monitored by the study team and descriptively compared between study arms.

SECONDARY OUTCOMES:
Incidence of community acquired respiratory viruses (CARV) | Up to 100 days post-transplant
  Will compare the cumulative incidence of CARV between study arms, counting death as a competing risk. Cox regression will be used to test for differences in the cause-specific hazard of CARV between study arms.
Frequency of respiratory viral symptoms | Up to 100 days post-transplant
  Will use Poisson generalized estimating equation regression models to compare the frequency of respiratory viral symptoms between study arms
Number of respiratory viral panel tests | Up to 100 days post-transplant
  Will compare the number of respiratory viral panel tests sent to the lab between study arms using Poisson regression with an offset for the number of days each participant was in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Pergam, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (2):
- United States (2):
  - University of Chicago Medicine-Orland Park, Orland Park, Illinois
  - Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2019-07-19): https://cdn.clinicaltrials.gov/large-docs/49/NCT04060849/ICF_000.pdf